CLINICAL TRIAL: NCT06670495
Title: Understanding the Human Papillomavirus Genotype Attribution and Disease Burden of Anal Cancer in China: A Multicenter Hospital-based Study
Brief Title: HPV Genotype Attribution and Disease Burden of Anal Cancer in China
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ying Zheng, Chief of Department, Fudan University
Other Study IDs: 2024-225-3778
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-08

CONDITIONS: Anal Cancer
Keywords: HPV prevalence; HPV genotype; Anal cancer
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — In this study, the qualified specimens will be obtained by biopsy, scraping, and swab for HPV DNA detection. Cancer tissue will be taken from patients with anal cancers. For surgical patients, cancer tissue can be obtained by biopsy or retrospective paraffin embedded tissue, for non-surgical patients, tissue can be obtained by biopsy. For tissue samples, cut about 5-25mg of the sample, put it into a 1.5ml centrifuge tube, add 180 Buffer AL and 20ul proteinase K solution, shake and mix well, centrifuge at low speed, and then store for testing. For retrospective paraffin embedded specimens, use a scalpel to remove excess paraffin and cut a 10um thick slice. If the surface of the specimen is exposed to air, discard the first 2-3 slices. Disassemble the microtome between blocks for decontamination.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To demonstrate HPV prevalence and its genotype distributions in anal cancer in China and to describe demographic and clinical features of HPV-related anal cancer in China; To describe the epidemiological characteristics ,trends and of disease burden of anal cancer in China

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients diagnosed with anal cancers, (2) Patients without radiation or chemotherapy prior to specimen collection;

Exclusion Criteria:

* (1) Patients with HIV infection, (2) Patients with immunosuppression after solid organ transplantation, (3) Those who do not agree to specimen collection and testing, (4) For retrospective study cases, those who without specimen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Patients with anal canal cancer: patients with anal canal cancer originating from the superior border of the functional anal canal (separated from the rectum) and defined as the palpable upper border of the anal sphincter and puborectalis muscles of the anorectal ring. It is approximately 3 to 5 cm in length, and its inferior border starts at the anal verge, the lowermost edge of the sphincter muscles, corresponding to the introitus of the anal orifice.
  2. Patients with perianal cancer: The perianal region starts at the anal verge and includes the perianal skin over a 5-cm radius from the squamous mucocutaneous junction
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence and types of distribution of HPV | From enrollment to pre-treatment
Incidence of anal-cancers-associated complications | From enrollment to pre-treatment
  with or without HPV infection by subgroups of sex, age at diagnosis, sexual orientation, and stage at diagnosis (Stage I, II, III, IV, unknown)
Routine laboratory testing results | From enrollment to pre-treatment

SECONDARY OUTCOMES:
Incidence rates of anal cancer in China | From enrollment to pre-treatment
  overall and for 5-year calendar periods 2001-2005, 2006-2010, and 2011-2015
Mortality rate of anal cancer in China | From enrollment to pre-treatment
  overall and for 5-year calendar periods 2001-2005, 2006-2010, and 2011-2015
Annual percentage changes (APCs) and average APCs (AAPCs) | From enrollment to pre-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No